CLINICAL TRIAL: NCT06802757
Title: A Phase II, Randomised, Open-label, Multicentre Study of Posaconazole Plus Pembrolizumab and Chemotherapy Versus Pembrolizumab and Chemotherapy as Neoadjuvant Therapy for Triple Negative Breast Cancer
Brief Title: Posaconazole Plus Pembrolizumab and Chemotherapy vs Pembrolizumab and Chemotherapy in Neoadjuvant Therapy for Triple Negative Breast Cancer
Acronym: PRISM-TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POS-PEM-Ⅱ-NEO-TNBC
Record Dates: First submitted 2025-01-16; First posted 2025-01-31 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Triple-Negative Breast Cancer; Pathological Complete Response; Neoadjuvant Therapy; Posaconazole
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — posaconazole; 130-nm albumin-bound paclitaxel; Carboplatin; Anthracyclines; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy + PD-1 inhibitor (Other): Nab-paclitaxel + carboplatin 4 cycles, sequential anthracycline + cyclophosphamide 4 cycles in combination with pembrolizumab
  Interventions: Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Anthracycline; Drug: Cyclophosphamide; Drug: Pembrolizumab
- Chemotherapy + PD-1 inhibitor+Posaconazole (Experimental): Nab-paclitaxel + carboplatin 4 cycles, sequential anthracycline + cyclophosphamide 4 cycles in combination with pembrolizumab and posaconazole
  Interventions: Drug: Posaconazole; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Anthracycline; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Posaconazole — Posaconazole 120mg/m2 po bid d1-14 q21d
  Arms: Chemotherapy + PD-1 inhibitor+Posaconazole
Drug: Nab-paclitaxel — Nab-paclitaxel 260mg/m2 d1 q21d
Drug: Carboplatin — Carboplatin AUC=6 d1 q21d
Drug: Anthracycline — Epirubicin 90-100mg/m2 d1 q21d or Doxorubicin 50-60mg/m2 d1 q21d
Drug: Cyclophosphamide — Cyclophosphamide 1000mg/m2 d1 q21d
Drug: Pembrolizumab — Pembrolizumab 200mg d1 q21d

SUMMARY:
Triple-negative breast cancer (TNBC) is as sociated with shorter overall survival than other breast cancer subtypes, despite the use of curative-intent anthracycline- and taxane-based systemic chemotherapy. Neoadjuvant therapy is now also recognized as the standard treatment for patients with high-risk TNBC. The Keynote-522 study demonstrated that the application of pembrolizumab has raised the pathological Complete Response (pCR) rate in TNBC to over 60%, but nearly 40% of patients still do not achieve pCR. How to further improve the pCR rate in TNBC patients has become a hot topic of current research.

Posaconazole is an antibiotic used to prevent invasive Aspergillus and Candida infections and to treat oropharyngeal candidiasis. Our preclinical studies have found that posaconazole can inhibit immune cell-mediated steroidogenesis to restrict TNBC tumor progression. The investigators design and begin a a prospective randomized controlled clinical study to explore the effectiveness of posaconazole in the neoadjuvant treatment of TNBC.

DETAILED DESCRIPTION:
OBJECTIVES: On the basis of chemotherapy combined with immunotherapy, posaconazole was used to further improve the pathological complete response (pCR) rate of high-risk triple-negative breast cancer (TNBC), and to explore biomarkers.

OUTLINE: From february 1st, 2025 to june 30th, 2026 the investigators will recruit 40 patients with first-time diagnosed early-stage TNBC. Enrolled patients were randomly divided into experimental group and control group on a 1:1 basis. Both groups received standard neoadjuvant chemotherapy combined with immunotherapy. The experimental group was treated with posaconazole (day 1: 300 mg po bid, from Day 2, start maintenance dose at 300 mg po qd, q21d). Standard surgical treatment was performed after 8 cycles and the surgical specimens were pathologically tested to compare the differences in pCR rates between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 and ≤ 70 years old;
2. first-confirmed TNBC;
3. cT1cN1-3M0 or cT2-4N0-3M0;
4. ECOG score 0-1 points.

Exclusion Criteria:

1. Stage I or IV;
2. History of previous breast cancer;
3. Patients with a history of other tumors who have received systemic therapy or local radiotherapy;
4. No immune system disease or connective tissue disease;
5. No history of hormone therapy;
6. Pregnant/lactating.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | 24 weeks
  Expected 10% increase in pCR rate

SECONDARY OUTCOMES:
Breast pathological complete response | 24 weeks
Objective response rate | 24 weeks
3-year event-free survival rate | After a median follow-up of 3 years
Survival rate | After a median follow-up of 3 years
Security | 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Center Shandong Cancer Hospital and Institute Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes